CLINICAL TRIAL: NCT02563223
Title: The Effect of Gravity on the Muscular Control of Landing From a Jump
Acronym: SLS-JUMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-118
Record Dates: First submitted 2015-07-23; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- electromyographic (EMG) measurements (Other): Interaction between gravity (weightlessness, hypergravity, and normal gravity) and pull-down force ont EMG amplitude and EMG timing.
  Interventions: Other: Parabolic flight; Device: Subject Loading System

INTERVENTIONS:
Other: Parabolic flight
Device: Subject Loading System — a device that combines a force platform on which the subject jumps and a Subject Loading System (SLS) that pulls the subject downwards.

SUMMARY:
In this project, investigators propose to study the jump in different reduced gravity fields obtained during parabolic flights profiles but also during increased gravity fields obtained during turns of the airplane or during the pull-up phase of the parabola. By means of a pneumatic device, an additional pull-down force will be added to the vertical force caused by the gravity field. By combining different levels of gravity to different levels of the added pull-down force it will be possible to dissociate the respective contribution of the otolithic and proprioceptive systems to the anticipatory landing response. To the investigators' knowledge, only one study has modified the gravity field during a jump. However, these authors did not add a pull-down force and only analyzed the vertical ground reaction force.

A better knowledge of the sensory-motor control of the landing phase of a jump will also increase the investigators' understanding of the physiopathology of joint instability. Indeed, similarities could be found between the evolution of the motor response due to the absence gravity during long-duration space flights and the pathological process of chronic ankle and knee instability. The knowledge generated by this study will thus provide invaluable information in the context of human performance and rehabilitation.

DETAILED DESCRIPTION:
Investigations description ----------------------------------

During the experiments, subjects will jump in different gravity fields while submitted to an additional pull-down force equal to 0-100% of their body weight on Earth. During the takeoff and landing phases of the jumps, the ground reaction force will be recorded by a force-platform, the movements of the limb segments will be recorded by means of a high-speed camera and the electrical activity (EMG) of the main lower limb muscles will be recorded by means of surface electrodes.

Force platform and Subject Loading System We have developed a device that combines a force platform on which the subject jumps and a Subject Loading System (SLS) that pulls the subject downwards.

The force platform is a 60 cm x 40 cm aluminum plate equipped with four force-transducers that measure the three components of the force exerted by the subject's feet on the ground.

The SLS consists in two pneumatic pistons, which are attached to a harness on one end and to the aluminum plate on the other. The SLS can be set to generate a force equal to 20-100% of the subject's body weight on Earth.

A security handrail (not shown on the picture) is attached to the aluminum plate, around the force-platform in case of unbalance of the subject.

EMG EMG will be recorded with a MyoSystem 1400L using surface electrodes. The skin will be shaved (if necessary) and the electrodes will be attached with double sided tape and plaster. The electrodes will be placed at the level of the lateral gastrocnemius, medial gastrocnemius, tibialis anterior and peroneus longus, and on the thigh at the level of the vastus lateralis, vastus medialis and lateral hamstrings and medial hamstrings. There will be 2 electrodes per muscle (fixed one against the other) and one reference electrode placed at the level of the C7 vertebra.

Manufacturer: Noraxon. Conformity certificate: CE 344

Video Movements of the subject will be recorded by means of a high-speed digital camera (Basler). In order to facilitate video analysis, 7 reflective markers (hemisphere with a 12 mm diameter) will delimit body segments: 3 will be glued on one shoe, 3 will be fixed on the skin (with the same method used for EMG electrodes) at the level of the ankle, knee, hip of one limb and the last one will be fixed on the neck.

Experimental protocol

----------------------------

Before flight subjects will be familiarized with the setup and the protocol. For each flight day, one subject will be studied. The procedure will be the following on all 3 days.

The experiment day starts at 7.30 a.m. with the test subject equipped with EMG electrodes and video markers. After take-off and after work is permitted, the subject goes to the experimental area where it is equipped with the SLS harness. Before each parabola, the subject stands beside the platform to adjust the zero level of the sensor (about 3 second). Then the subject steps on the platform to record his weight (about 3 second).

During the hypergravity initial part in of the parabola, the subject is standing with is two feet on each side of the platform. The traction system is loose (5 kg traction). During the injection, the traction system starts to progressively pull downwards on the subject. The traction force is tuned between 20% and 100% of body weight on Earth. The traction force is constant during each parabola. During the 20 second of weightlessness or partial gravity, the subject jumps several times. At the end of the parabola, the subject puts his feet at the side of the platform and the traction system stops to pull downwards before the pull out phase.

This experiment will also be performed during periods of increased gravity obtained during turns of the airplane. Three turns per flight should be performed at 3 levels of gravity: 1.2, 1.4 g and 1.6 g.

During each parabola or turn, one experimenter is taking care of the control of the traction system and of the collection of the data, a second one takes care of the image acquisition, and a third one takes care of the modification of the configuration of the harness between the parabolas and of the safety of the subject in case of unbalance during the parabolas or during the turn.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude. There will be no additional test performed for subject selection

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women
* Person with medical history of musculoskeletal disorders of the lower limbs, pelvis or spine, neurological or vestibular disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Electromyography (Amplitude - mV and latency - ms) | baseline
  EMG (electrical activity produced my muscles when they contract) will be recorded with a MyoSystem 1400L using surface electrodes at the level of the lateral gastrocnemius, medial gastrocnemius, tibialis anterior and peroneus longus, and on the thigh at the level of the vastus lateralis, vastus medialis and lateral hamstrings and medial hamstrings.
  EMG activation (amplitude and latency) will be measured during jumps at different level of gravity and pull-down forces.

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France